CLINICAL TRIAL: NCT06255691
Title: 10-year Follow-up After 24/7-phone Support After Aortic Valve Replacement Surgery in Early Rehabilitation Study
Brief Title: 10-year Follow-up After Aortic Valve Replacement Surgery
Acronym: AVR-10year
Status: Not yet recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Stein Ove Danielsen, Associate professor, Oslo University Hospital
Other Study IDs: 23596
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Aortic Stenosis; Anxiety; Depressive Symptoms; Quality of Life
Keywords: aortic valve replacement; longitudinal study; patient reported outcome; symptoms of anxiety; health-related quality of life
MeSH Terms: conditions — Aortic Valve Stenosis; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is a lack of data on patients self-reported outcomes (PROMs) on health-related quality of life (HRQoL)and symptoms on anxiety and depression 10 years after Surgical After Aortic Valve Replacement (SAVR), and patient reported experiences with the health services (PREMS). In this 10-years follow-up study on patients alive from the study named "The Impact of 24/ 7-phone Support on Readmission After Aortic Valve Replacement, a Randomized Clinical Trial (AVRre)" NCT02522663 we will repeat the survey on symtoms on anxiety and depresion using Hospital Anxiety and depression Scale (HADS), health-related quality of life (EQ-5D) and questions about experiences with the health services.

DETAILED DESCRIPTION:
"The Impact of 24/ 7-phone Support on Readmission After Aortic Valve Replacement, a Randomized Clinical Trial (AVRre) was a prospective, randomized controlled study (RSC) Including 286 patients after AVR from 2015 til 2017, NCT02522663. The results reported in international publications showed reduced symptoms on anxiety the first month after AVR.

Reduction of anxiety revealed to be an important aim for the intervention. We found that symptoms of anxiety in the early rehabilitation phase after discharge following surgical aortic valve replacement phase was significantly reduced.

There is a lack of data on patients self-reported outcome on symptoms on anxiety and depression 10 years after Surgical After Aortic Valve Replacement (SAVR), and patient reported experiences with health services. In this 10-years follow-up study on patients alive from the study named "The Impact of 24/ 7-phone Support on Readmission After Aortic Valve Replacement, a Randomized Clinical Trial (AVRre)" NCT02522663 we will conduct a survey on symtoms of anxiety and depresion using Hospital Anxiety and depression Scale (HADS), quality of life (EQ-5D) and questions about experiences with health services.

The results of the planned 10-years follow-up may give guidance in how to allocate health resources and planning for and follow-up of patients after heart surgery.

ELIGIBILITY:
Inclusion Criteria:

Treatment with AVR (biological or mechanical) single, AVR (b or m)+aortocoronary bypass, AVR (b or m)+supra coronary tube graft Can understand, speak and write native Language (norwegian), and be able to fill in the questionnaires

-

Exclusion Criteria:

Patients not alive after the AVRre study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 year follow-up of the participants in the AVrRe study
Sampling Method: Non-Probability Sample
Enrollment: 282 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Symptoms of anxiety and depression | 10 year follow-up
  Symptoms of anxiety and depression measured by Hospital Anxiety and Depression Scale (HADS)
Health related quality of life | 10 year follow-up
  EQ-5D-3L questionnaire from The EuroQol Group to measure health related quality of life.

SECONDARY OUTCOMES:
Experiences with health services | 10 year follow-up
  Open questions

CONTACTS AND LOCATIONS:
Overall Officials: Stein Ove O Danielsen, PhD, Principal Investigator — OsloMet